CLINICAL TRIAL: NCT03047590
Title: Comparison of Affect-based, Self-selected, and Traditional Exercise Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Zachary, Postdoctoral Associate, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D0991
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity
Keywords: exercise behavior; exercise prescription; affect-based exercise; affect-guided exercise; self-paced exercise; self-selected exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Choice-No Affect (Experimental): These participants self-select (i.e., choose) their exercise intensity with the goal of walking 30-60 minutes on most days of the week. For safety reasons, they are instructed not to exceed 59% of their heart rate reserve. This is choice-based exercise intensity with no focus on positive affect.
  Interventions: Behavioral: Choice-based Exercise Intensity
- Choice-Affect (Experimental): These participants self-select their exercise intensity with the goal of walking 30-60 minutes on most days of the week. They're instructed to choose the intensity that makes them feel the best. For safety reasons, they are instructed not to exceed 59% of their heart rate reserve. This is choice-based exercise intensity with a focus on positive affect.
  Interventions: Behavioral: Choice-based Exercise Intensity; Behavioral: Positive Affect Focus
- No Choice-Affect (Experimental): These participants regulate their exercise intensity using their heart rate, with the goal of walking 30-60 minutes on most days of the week. The intensity is "moderate" according to the American College of Sports Medicine (40-59% of their heart rate reserve). Meanwhile, these participants are instructed to focus on the "good feelings" that come with exercise. this is heart rate-based exercise intensity with a focus on positive affect.
  Interventions: Behavioral: Positive Affect Focus; Behavioral: Heart rate-based Exercise Intensity
- No Choice-No Affect (Active Comparator): These participants regulate their exercise intensity using their heart rate, with the goal of walking 30-60 minutes on most days of the week. The intensity is "moderate" according to the American College of Sports Medicine (40-59% of their heart rate reserve). This is heart rate-based exercise intensity with no focus on positive affect.
  Interventions: Behavioral: Heart rate-based Exercise Intensity

INTERVENTIONS:
Behavioral: Choice-based Exercise Intensity — Participants are instructed to choose whichever intensity they want, rather than regulate their intensity based on heart rate.
  Arms: Choice-Affect; Choice-No Affect
Behavioral: Positive Affect Focus — Participants are instructed to focus on feeling good while exercising.
  Arms: Choice-Affect; No Choice-Affect
Behavioral: Heart rate-based Exercise Intensity — Participants are instructed to regulate their exercise intensity based on their heart rate.
  Arms: No Choice-Affect; No Choice-No Affect

SUMMARY:
This study will evaluate adherence to four types of walking programs. Participants will be randomized to walking programs that included either (1) affect-based exercise intensity, (2) self-selected (or "choice-based") exercise intensity, (3) heart-rate based exercise intensity, or (4) heart-rate guided exercise intensity with the emphasis on affective benefits.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an "affect-based" or "choice-based" exercise prescription is more effective for behavior change than a traditional, "moderate-intensity" exercise prescription. Prior research suggests that "choice-based" or "self-selected" exercise intensity is more pleasant and adhered to than "moderate-intensity exercise" (Williams et al., 2014). Similarly, affect-based exercise prescriptions (i.e., an exercise prescription where intensity is regulated based on the pleasure-displeasure one feels while exercising) appear to have merit (Baldwin, Kangas, Denman, Smits, Yamada, & Otto, 2016).

However, choice-based and affect-based exercise prescriptions have not been compared to each other. Further, it is unknown if it is the intensity regulation that matters (e.g., "choose an intensity that feels good" or the focus on affect (e.g., "focus on feeling good). Third, prior research has not objectively measured physical activity behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be fluent in English
* Must be able to walk
* Exercise less than 90 minutes per week at a moderate-intensity
* Must be able to attend laboratory visits
* Must have mobile internet accent and a personal smartphone (iPhone iOS 9+ or Android OS 4.3+)
* Can safely exercise at an intensity that is at least "moderate"

Exclusion Criteria:

* People who are recommended to have medical clearance prior to exercising, according to the American College of Sports Medicine's preparticipation screening criteria, will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured exercise behavior | This will be measured throughout the baseline assessment period (2 weeks) and intervention period (4 weeks)
  Minutes per week of objectively measured exercise behavior.

SECONDARY OUTCOMES:
Change in self-reported exercise behavior | This will be measured throughout the baseline assessment period (2 weeks) and intervention period (4 weeks)
  Minutes per week of self-reported exercise behavior that is reported using exercise log.
Change in affective attitudes | Measured during baseline assessment period and at the end of the intervention
  Affective attitudes toward exercise
Self-reported intrinsic motivation (questionnaires) | Two weeks into study intervention
  Intrinsic motivation for exercise program
Enjoyment | Measured at the end of the intervention period (4 weeks)
  Enjoyment of exercise program.
Change in weight | Measured at the beginning and end of the study (6 weeks).
  Body weight
Change in resting heart rate | Measured at the beginning and end of the study (6 weeks).
  Resting heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University IBRC Lab, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators retain ownership of all study data, but are willing to share anonymized data for transparency purposes at the conclusion of the study. Data may be requested by contacting the Principal Investigator.

REFERENCES:
- [Background] Baldwin AS, Kangas JL, Denman DC, Smits JA, Yamada T, Otto MW. Cardiorespiratory fitness moderates the effect of an affect-guided physical activity prescription: a pilot randomized controlled trial. Cogn Behav Ther. 2016 Nov;45(6):445-57. doi: 10.1080/16506073.2016.1194454. Epub 2016 Jun 16. PMID 27310568
- [Background] Williams DM, Dunsiger S, Miranda R Jr, Gwaltney CJ, Emerson JA, Monti PM, Parisi AF. Recommending self-paced exercise among overweight and obese adults: a randomized pilot study. Ann Behav Med. 2015 Apr;49(2):280-5. doi: 10.1007/s12160-014-9642-7. PMID 25223963